CLINICAL TRIAL: NCT03189589
Title: A Randomised, Double-blind, Parallel Group Study to Evaluate the Safety, Tolerability and Pharmacokinetics of a Single Dose of GSK2269557 Administered Via the ELLIPTA™ Dry Powder Inhaler to Healthy Participants
Brief Title: Safety, Tolerability and Pharmacokinetics (PK) Study of GSK2269557 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207674; 2017-001073-16 (EudraCT Number)
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Results first posted 2019-01-14 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pharmacokinetics; Healthy; ELLIPTA; Safety; GSK2269557; Inhalation; Tolerability
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Nemiralisib

STUDY DESIGN:
Intervention Model Description: Healthy subjects will be randomized to receive GSK2269557 750 µg or GSK2269557 500 µg.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study and subjects and investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK2269557 500 µg receivers (Experimental): Randomized healthy subjects will receive single dose of GSK2269557 500 µg via inhalation route via the ELLIPTA DPI.
  Interventions: Drug: GSK2269557 500 µg
- GSK2269557 750 µg receivers (Experimental): Randomized healthy subjects will receive single dose of GSK2269557 750 µg via inhalation route via the ELLIPTA DPI.
  Interventions: Drug: GSK2269557 750 µg

INTERVENTIONS:
Drug: GSK2269557 500 µg — GSK2269557 is a potent and highly selective inhaled Phosphoinositide 3 Kinase delta inhibitor. Single dose of GSK2269557 500 µg will be administered to randomized subjects via inhalation route using ELLIPTA DPI.
  Arms: GSK2269557 500 µg receivers
Drug: GSK2269557 750 µg — GSK2269557 is a potent and highly selective inhaled Phosphoinositide 3 Kinase delta inhibitor. Single dose of GSK2269557 750 µg will be administered to randomized subjects via inhalation route using ELLIPTA DPI.
  Arms: GSK2269557 750 µg receivers

SUMMARY:
GSK2269557 is being developed as an anti-inflammatory and anti-infective agent for the treatment of inflammatory airways diseases. This is the first study using a new formulation of GSK2269557 in healthy subjects and will evaluate the safety, tolerability and PK of a single dose of GSK2269557. Data derived from this study will inform on the PK profile and systemic exposure expected during Phase 2b. Approximately twelve healthy subjects will be randomized to receive a single dose of GSK2269557 750 micrograms (µg) or a single dose of GSK2269557 500 µg via the ELLIPTA® dry powder inhaler (DPI) formulated in a blend containing 0.4 percent magnesium stearate (MgSt) in 1:1 ratio. This randomized, parallel group study will be carried out in 3 phases, including screening phase, treatment phase and follow-up phase. The total study duration for each subject will be up to 6 weeks. ELLIPTA is a registered trademark of GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 75 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG tests. Re-screening will be allowed once, at the discretion of the Principal Investigator in consultation with GlaxoSmithKline (GSK) medical monitor.
* Normal spirometry at Screening FEV1 and FVC >=80 percent of predicted (measurements to be taken in triplicate and the highest value for each component must be >=80 percent of predicted).
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 18.0 - 35.0 kg per square meter (kg/m^2) (inclusive).
* Male or female: A male subject must agree to use contraception during the treatment period for at least 5 half-lives plus 90 days after the last dose of study treatment and refrain from donating sperm during this period. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or A WOCBP who agrees to follow the contraceptive guidance during the treatment period for at least 5 half-lives plus 90 days after the last dose of study treatment.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Asthma or a history of asthma (except in childhood, which has now remitted).
* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Abnormal blood pressure [as determined by the investigator].
* Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTc interval >450 milliseconds (msec).
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing.
* Live vaccine(s) within 1 month prior to screening, or plans to receive such vaccines during the study.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) within 56 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day. Consider adding the following criteria if subjects can only be enrolled once per study.
* Current enrollment or past participation within the last 90 days before signing of consent in any other clinical study involving an investigational study treatment or any other type of medical research
* Presence of Hepatitis B surface antigen (HBsAg) at screening Positive Hepatitis C antibody test result at screening. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C Ribonucleic Acid (RNA) test is obtained.
* Positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 3 months prior to the study defined as: An average weekly intake of >14 units for males and females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current smoker or a history of smoking within 6 months of Screening, or a total pack year history of >5 pack years. [Number of pack years = (number of cigarettes per day/20) multiplied by number of years smoked]
* Sensitivity to any of the study treatments, or components thereof (including lactose and MgSt), or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=207674

REFERENCES:
- [Background] Wilson R, Templeton A, Leemereise C, Eames R, Banham-Hall E, Hessel EM, Cahn A. Safety, Tolerability, and Pharmacokinetics of a New Formulation of Nemiralisib Administered via a Dry Powder Inhaler to Healthy Individuals. Clin Ther. 2019 Jun;41(6):1214-1220. doi: 10.1016/j.clinthera.2019.04.008. Epub 2019 May 7. PMID 31076203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in the United Kingdom from 15-June-2017 to 24-July-2017.
Pre-assignment Details: A total of 19 participants were screened for this study, of which 7 participants were screen failures and 12 participants were randomized to treatment. The reasons for screen failure were: did not meet inclusion/exclusion criteria (6 participants) and withdrawal by participant (1 participant).
Groups:
- GSK2269557 500 mcg: Eligible participants received a single dose of GSK2269557 500 micrograms (mcg) via the ELLIPTA dry powder inhaler (DPI) on Day 1.
- GSK2269557 750 mcg: Eligible participants received a single dose of GSK2269557 750 mcg via the ELLIPTA DPI on Day 1.
Period: Overall Study
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK2269557 500 mcg: Eligible participants received a single dose of GSK2269557 500 mcg via the ELLIPTA DPI on Day 1.
- Total: Total of all reporting groups
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (6.21) | 42.7 (10.98) | 48.3 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean GSK2269557 Plasma Concentration
Description: Whole blood samples of approximately 2 milliliters were collected for measurement of plasma concentrations of GSK2269557 at the indicated time points. The pharmacokinetic parameters were calculated by standard non-compartmental analysis. Pharmacokinetic (PK) Population which comprised of all randomized participants in the Safety Population and for whom a PK sample was obtained and analyzed.
Time Frame: Day 1: Pre-dose, 5 minutes post dose, 30 minutes post-dose, 2 hours post-dose, 6 hours post-dose, 12 hours post-dose; Day 2: 24 hours post-dose; Day 3: 48 hours post-dose and Day 6: 120 hours post-dose
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Picograms per milliliter
  Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  5 minutes post-dose | 2175.5 (843.68) | 1871.8 (985.15)
  30 minutes post-dose | 480.7 (155.28) | 530.7 (260.82)
  2 hours post-dose | 322.9 (83.85) | 414.6 (187.63)
  6 hours post-dose | 259.7 (81.60) | 424.0 (186.51)
  12 hours post-dose | 210.5 (52.94) | 319.5 (109.94)
  24 hours post-dose | 171.8 (48.71) | 248.9 (71.92)
  48 hours post-dose | 114.0 (38.31) | 145.2 (40.54)
  120 hours post-dose | 36.3 (19.30) | 40.1 (26.37)

2. Primary Outcome: Area Under the Plasma Drug Concentration Versus Time Curve (AUC) From Zero to Time t (AUC [0 to t]), AUC From Zero to 24 Hours (AUC [0 to 24]) and AUC From Zero to Infinity (AUC [0 to Inf]) of GSK2269557
Description: Blood samples were collected to evaluate the PK of GSK2269557 at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis. Only those participants with data available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours*picograms per milliliter
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Hours*picograms per milliliter
  AUC (0 to t), n=6,6 | 14032.8 (5027.09) | 18468.7 (7007.72)
  AUC (0 to 24), n=6,6 | 6000.6 (1646.07) | 8497.7 (3189.43)
  AUC (0 to inf), n=4,5: number analyzed (Participants) | 4 | 5
  AUC (0 to inf), n=4,5 | 19291.7 (3788.10) | 23340.9 (6395.14)

3. Primary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) and Concentration at Trough (Ctrough) of GSK2269557
Description: Blood samples were collected to evaluate the PK of GSK2269557 at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Picograms per milliliter
  Cmax | 2175.5 (843.68) | 1871.8 (985.15)
  Ctrough | 171.8 (48.71) | 248.9 (71.92)

4. Primary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax) and Terminal Half-life (t1/2)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Hours
  Tmax, n=6,6 | 0.083 [0.08 to 0.10] | 0.083 [0.07 to 0.083]
  t1/2, n=4,5: number analyzed (Participants) | 4 | 5
  t1/2, n=4,5 | 42.7 [42 to 48] | 38.2 [31 to 49]

5. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Vital signs included blood pressure (systolic and diastolic blood pressure) and heart rate measurements and were assessed with the participant in a semi-supine position after 5 minutes rest. The potential clinical concern range values for vital signs were: systolic blood pressure (lower <85 millimeters of mercury and higher >160 millimeters of mercury), diastolic blood pressure (lower <45 millimeters of mercury and higher >100 millimeters of mercury) and heart rate (lower <40 beats per minute and higher >110 beats per minute). Number of participants with vital signs of potential clinical importance are presented. Safety Population comprised of all randomized participants who received at least one dose of study treatment.
Time Frame: Up to Day 2
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Importance
Description: Twelve-lead ECG was obtained using an ECG machine which automatically measured PR, QRS, QT and corrected QT (QTc) intervals. ECG parameters and their potential clinical importance range values were: absolute QTc interval (lower >450 milliseconds [msec]), absolute PR interval (lower <110 msec and upper >220 msec), absolute QRS interval (lower <75 msec and upper >110 msec). Number of participants with electrocardiogram (ECG) values of potential clinical importance are presented.
Time Frame: Up to Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

7. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 Second (FEV1)
Description: The maximal amount of air forcefully exhaled in 1 second (FEV1) and forced vital capacity (FVC) was measured using a spirometer. Baseline was latest pre-dose assessment. Change from Baseline was calculated by subtracting Baseline values from post-dose visit values. Mean change from Baseline in FVC and FEV1 is presented.
Time Frame: Baseline and Day 1
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Liters (L)
  FEV1 | 0.027 (0.0554) | -0.040 (0.2060)
  FVC | 0.177 (0.0836) | 0.065 (0.2780)

8. Secondary Outcome: Number of Participants With Hematology Abnormalities of Potential Clinical Importance
Description: Hematology parameters and their potential clinical concern values were: Hematocrit (high flag: >0.54 and change from Baseline: decrease of 0.075), hemoglobin (high flag: >180 grams per Liter and change from Baseline: decrease of 25 grams per Liter), lymphocytes (low flag: <0.8*10^9 cells per Liter), neutrophil count (low flag: <1.5*10^9 cells per Liter), platelet count (low flag: <100*10^9 cells per Liter and high flag: >550*10^9 cells per Liter) and white blood cell count (low flag: <3*10^9 cells per Liter and high flag: >20*10^9 cells per Liter). Number of participants with hematology abnormalities of potential clinical importance are presented.
Time Frame: Up to Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance
Description: Clinical chemistry parameters and their potential clinical concern range values were: calcium (low flag <2 millimoles/Liter [mmol/L] and high flag >2.75 mmol/L), creatinine (high flag >44.2 micromoles/Liter increase in change from Baseline), glucose (fasting) (<3 mmol/L and >9 mmol/L), potassium (low flag <3 mmol/L and high flag >5.5 mmol/L above ULN), sodium (low flag <130 mmol/L and high flag >150 mmol/L). Number of participants with clinical chemistry abnormalities of potential clinical importance are presented.
Time Frame: Up to Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 12 days post-dose
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
Number analyzed (Participants) | 6 | 6
Participants
  AE | 3 | 3
  SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 days post-dose
Description: AE and SAE were collected for the Safety Population which comprised of all randomized participants who received at least one dose of study treatment.
Arm/Group | GSK2269557 500 mcg | GSK2269557 750 mcg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2269557 500 mcg (N=6) | GSK2269557 750 mcg (N=6)
Fatigue (General disorders) | 0 (0) | 2 (2)
Catheter site inflammation (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03189589/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT03189589/SAP_001.pdf